CLINICAL TRIAL: NCT04660188
Title: Impact of a Breast cAncer Survivorship Interprofessional Community Care Model (BASIC): A Randomized Controlled Trial
Brief Title: Impact of a Breast cAncer Survivorship Interprofessional Community Care Model
Acronym: BASIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National University of Singapore (Other); SingHealth Polyclinics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/2452
Record Dates: First submitted 2020-03-18; First posted 2020-12-09 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Survivorship; Breast Cancer
Keywords: survivorship care model; breast cancer survivor; shared-care; primary care; interprofessional; cancer survivorship
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary collaborative care arm (Experimental): Post-treatment clinical follow-up visits will be staggered between the oncologist and a dedicated PCP. A patient navigator will be assigned to each study participant to conduct follow-up sessions over the phone regularly at an approximate interval of 3 months.
  Interventions: Other: Multidisciplinary collaborative care arm
- Attentional control arm (No Intervention): BCS will receive follow-up care by their oncologists and any other healthcare providers under existing usual care practices at NCCS.

INTERVENTIONS:
Other: Multidisciplinary collaborative care arm — Study participants will be cared for by a team of healthcare professionals; an oncologist, a PCP and a pharmacist navigator.
  Arms: Multidisciplinary collaborative care arm

SUMMARY:
With an increase in breast cancer survivors (BCS) in Singapore, the current oncologist-centric survivorship model will not be sustainable to respond to the rising demand of survivorship care services. To meet the long-term healthcare needs of Singaporeans in a sustainable manner, the investigators propose to pilot a breast cancer survivorship inter-professional community (BASIC) care model for cancer survivorship. This pilot study aims to assess the feasibility and acceptability of this care model for implementation among BCS and healthcare providers. The investigators hypothesize that the BASIC model is feasible and acceptable to be evaluated on a larger scale. This new follow-up model can potentially reduce waiting times in tertiary centers without compromising quality of care, directly benefiting participants through more efficient follow-up sessions.

DETAILED DESCRIPTION:
In Singapore, breast cancer accounts for approximately 30% of all new cancer cases. With an overall 10-year age-standardized survival rate of 50%, it is estimated that 900 BCS will require dedicated cancer survivorship care in Singapore annually. However, the current oncologist-centric survivorship model adopted in Singapore will not be sustainable to respond to the rising demand for survivorship care services. This inability to cope with the growing demand poses a major challenge to the health system and accentuates an emerging need for an alternative evidence-based care model to support BCS and healthcare providers in achieving efficient and effective cancer survivorship care.

The American Society of Clinical Oncology (ASCO) advocates a collaborative survivorship care model involving the transition of cancer survivors from specialist to primary care setting via a risk-stratified approach. While the proposed collaborative model is promising and appealing, its feasibility and applicability in the local Asian setting considering cultural and socioeconomic factors is unknown. Furthermore, two major gaps exist: (i) there is a lack of comprehensive evaluation of structural factors in care coordination and clinical outcomes determination; and (ii) the potential of community pharmacists in cancer survivorship care is not maximized.

The main objective of the study is to assess the feasibility and acceptability of the BASIC care model for implementation amongst BCS and healthcare providers. The secondary objective addresses the effectiveness of BASIC model by providing robust parameters estimation for the physical symptom distress burden and quality of life outcome measures that will be used for sample size calculation in the eventual main trial.

This will be a pragmatic, randomized, controlled, pilot trial conducted at the National Cancer Centre Singapore (NCCS), participating SingHealth polyclinics and Watsons community pharmacies over a period of 2 years. Participants will be randomized into the multidisciplinary collaborative care arm or attentional control arm in a 1:1 ratio, stratified by the absence versus presence of comorbidities. In the multidisciplinary collaborative care arm, participants will experience a 12-month cancer follow-up schedule via a shared-care approach. In the attentional control arm, participants will continue with usual care.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older.
* Received a formal diagnosis of breast cancer.
* At least three years after active primary treatment including surgery, chemotherapy, radiotherapy (if any) and targeted therapy (if any).
* Ascertained to be a low-risk cancer survivor by oncologist.
* Ambulatory with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, indicative of adequate functioning capacity to travel and receive follow-up care at polyclinics.
* Able to read and understand either English or Mandarin

Exclusion Criteria:

* Physically or mentally incapable of providing verbal/ written consent.
* Unwell or unable to comply with the study protocol that involves questionnaires completion.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer survivors
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in participants' health-related quality of life | Baseline, every 3 months up to 12 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) is used. The EORTC QLQ-C30 consists of five functional scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, nausea/ vomiting and pain), a global quality of life status and six single item measures (dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial stability). All scales are scored from 0 to 100 where a higher score on functioning and global health status scales is indicative of better functioning; and a higher score on symptom scales and single items is indicative of a higher symptom burden.
Change in participants' physical and psychological symptom distress levels | Baseline, every 3 months up to 12 months
  The Rotterdam Symptom Checklist (RSCL) is used. The physical domain of the RSCL comprises of 23 items and the psychological distress domain comprises of 7 items. Each item will be rated on a 4-point Likert scale ("not at all", "a little", "quite a bit" and "very much"). A total physical symptom distress score can be summed to give a final score between 23 to 92, where a higher score indicates a higher symptom distress level. A total psychological distress score can be summed to give a final score between 7 to 28, where a higher score indicates a higher psychological distress level.

SECONDARY OUTCOMES:
Participants' satisfaction with the shared-care model | One year post-intervention
  Participants in the intervention arm who received the intervention will complete an overall satisfaction questionnaire. This questionnaire is adapted from Patient Experience Measures from the CAHPS Cancer Care Survey. It comprises of 21 items divided into 4 sections evaluating (1) care accessibility and adequacy (8 items); (2) overall communication (5 items); (3) care coordination (3 items); and (4) satisfaction with care (5 items). 20 items will be rated on a Likert scale, where a higher score indicating better experience and satisfaction. One item is an open response question for participants' feedback.
Change in participants' health utilities | Baseline, every 3 months up to 12 months
  The EuroQol 5-Dimensions (EQ-5D-5L) has five dimensions: mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. Each dimension will be rated on a 5-point Likert scale ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems"), where a higher score indicating greater severity. The second part consists of a visual analogue scale ranging from 0 (worst health imagined) to 100 (best health imagined) where participants will mark on the scale and write down the corresponding number to indicate their health state. Results from the EQ-5D-5L will be used to derive preference-based measures of health-related quality of life to estimate health utilities.
Change in healthcare cost and productivity | Baseline, every 6 months up to 12 months
  A healthcare utilization survey is used where open-ended questions require participants to report their expenditure to outpatient clinics, hospitalization episodes and on medication. The second part gathers information on the work-related outcomes including change in job scope, paid/ unpaid leave and change in productivity.
Rate of adherence to breast cancer survivorship care guidelines | From start to end of study, up to 12 months
  The rate of adherence to evidence-based breast cancer survivorship care guidelines will be determined by the proportion of participants who satisfied each of the following areas based on documentation of review or scans/ procedures ordered: (1) annual mammograms; (2) screening for secondary primary cancers; (3) assessment and management of physical and psychosocial long-term and late effects of breast cancer or treatment; (4) health promotion; and (5) care coordination.

CONTACTS AND LOCATIONS:
Overall Officials: Rose WY Fok, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halpern MT, Viswanathan M, Evans TS, Birken SA, Basch E, Mayer DK. Models of Cancer Survivorship Care: Overview and Summary of Current Evidence. J Oncol Pract. 2015 Jan;11(1):e19-27. doi: 10.1200/JOP.2014.001403. Epub 2014 Sep 9. PMID 25205779
- [Background] Grunfeld E, Fitzpatrick R, Mant D, Yudkin P, Adewuyi-Dalton R, Stewart J, Cole D, Vessey M. Comparison of breast cancer patient satisfaction with follow-up in primary care versus specialist care: results from a randomized controlled trial. Br J Gen Pract. 1999 Sep;49(446):705-10. PMID 10756611
- [Background] Grunfeld E, Levine MN, Julian JA, Coyle D, Szechtman B, Mirsky D, Verma S, Dent S, Sawka C, Pritchard KI, Ginsburg D, Wood M, Whelan T. Randomized trial of long-term follow-up for early-stage breast cancer: a comparison of family physician versus specialist care. J Clin Oncol. 2006 Feb 20;24(6):848-55. doi: 10.1200/JCO.2005.03.2235. Epub 2006 Jan 17. PMID 16418496
- [Background] Blaauwbroek R, Tuinier W, Meyboom-de Jong B, Kamps WA, Postma A. Shared care by paediatric oncologists and family doctors for long-term follow-up of adult childhood cancer survivors: a pilot study. Lancet Oncol. 2008 Mar;9(3):232-8. doi: 10.1016/S1470-2045(08)70034-2. Epub 2008 Feb 20. PMID 18282804
- [Background] Ke Y, Ng T, Chan A. Survivorship care models for breast cancer, colorectal cancer, and adolescent and young adult (AYA) cancer survivors: a systematic review. Support Care Cancer. 2018 Jul;26(7):2125-2141. doi: 10.1007/s00520-018-4197-y. Epub 2018 Apr 25. PMID 29696424
- [Background] Ng T, Toh MR, Cheung YT, Chan A. Follow-up care practices and barriers to breast cancer survivorship: perspectives from Asian oncology practitioners. Support Care Cancer. 2015 Nov;23(11):3193-200. doi: 10.1007/s00520-015-2700-2. Epub 2015 Mar 21. PMID 25791392
- [Background] Chan A, Lum ZK, Ng T, Eyob T, Wang XJ, Chae JW, Dorajoo S, Shwe M, Gan YX, Fok R, Loh KW, Tan YP, Fan G. Perceptions and Barriers of Survivorship Care in Asia: Perceptions From Asian Breast Cancer Survivors. J Glob Oncol. 2016 Jun 8;3(2):98-104. doi: 10.1200/JGO.2016.004929. eCollection 2017 Apr. PMID 28717749
- [Background] Chan A, Gan YX, Oh SK, Ng T, Shwe M, Chan R, Ng R, Goh B, Tan YP, Fan G. A culturally adapted survivorship programme for Asian early stage breast cancer patients in Singapore: A randomized, controlled trial. Psychooncology. 2017 Oct;26(10):1654-1659. doi: 10.1002/pon.4357. Epub 2017 Jan 25. PMID 28024163
- [Background] Lim HA, Mahendran R, Chua J, Peh CX, Lim SE, Kua EH. The Distress Thermometer as an ultra-short screening tool: a first validation study for mixed-cancer outpatients in Singapore. Compr Psychiatry. 2014 May;55(4):1055-62. doi: 10.1016/j.comppsych.2014.01.008. Epub 2014 Jan 18. PMID 24556515
- [Background] Breitenstein SM, Gross D, Garvey CA, Hill C, Fogg L, Resnick B. Implementation fidelity in community-based interventions. Res Nurs Health. 2010 Apr;33(2):164-73. doi: 10.1002/nur.20373. PMID 20198637
- [Background] van Onzenoort HA, Menger FE, Neef C, Verberk WJ, Kroon AA, de Leeuw PW, van der Kuy PH. Participation in a clinical trial enhances adherence and persistence to treatment: a retrospective cohort study. Hypertension. 2011 Oct;58(4):573-8. doi: 10.1161/HYPERTENSIONAHA.111.171074. Epub 2011 Aug 8. PMID 21825228
- [Background] Gao F, Ng GY, Cheung YB, Thumboo J, Pang G, Koo WH, Sethi VK, Wee J, Goh C. The Singaporean English and Chinese versions of the EQ-5D achieved measurement equivalence in cancer patients. J Clin Epidemiol. 2009 Feb;62(2):206-13. doi: 10.1016/j.jclinepi.2008.03.007. Epub 2008 Jul 10. PMID 18619790
- [Background] Cheung YB, Thumboo J, Goh C, Khoo KS, Che W, Wee J. The equivalence and difference between the English and Chinese versions of two major, cancer-specific, health-related quality-of-life questionnaires. Cancer. 2004 Dec 15;101(12):2874-80. doi: 10.1002/cncr.20681. PMID 15529310
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Tan ML, Idris DB, Teo LW, Loh SY, Seow GC, Chia YY, Tin AS. Validation of EORTC QLQ-C30 and QLQ-BR23 questionnaires in the measurement of quality of life of breast cancer patients in Singapore. Asia Pac J Oncol Nurs. 2014 Apr-Jun;1(1):22-32. doi: 10.4103/2347-5625.135817. PMID 27981079
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Ng T, Dorajoo SR, Cheung YT, Lam YC, Yeo HL, Shwe M, Gan YX, Foo KM, Loh WK, Koo SL, Jain A, Lee GE, Dent R, Yap YS, Ng R, Chan A. Distinct and heterogeneous trajectories of self-perceived cognitive impairment among Asian breast cancer survivors. Psychooncology. 2018 Apr;27(4):1185-1192. doi: 10.1002/pon.4635. Epub 2018 Feb 1. PMID 29315963
- See also: Singapore Cancer Registry: Annual Registry Report 2015 — https://www.nrdo.gov.sg/docs/librariesprovider3/Publications-Cancer/cancer-registry-annual-report-2015_web.pdf?sfvrsn=10
- See also: Speech by Minister of State for Health, Dr Lam Pin Min, at the MOH Committee of Supply debate 2017 — https://www.moh.gov.sg/news-highlights/details/speech-by-minister-of-state-for-health-dr-lam-pin-min-at-the-moh-committee-of-supply-debate-2017
- See also: Sympton burden and medication use in adult sarcoma patients — https://link.springer.com/article/10.1007/s00520-014-2533-4